CLINICAL TRIAL: NCT05743881
Title: A Phase 1, Randomized, Observer-blind, Placebo-controlled, Age De-escalation Study of the Safety, Tolerability, and Immunogenicity of mRNA-1345 and mRNA-1365 in Participants Aged 5 Months to <24 Months
Brief Title: A Safety, Tolerability, and Immunogenicity Study of mRNA-1345 and mRNA-1365 in Participants Aged 5 Months to <24 Months
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: mRNA-1365-P101; 2022-502022-41 (EudraCT Number); 2022-502022-41-00 (Other: EU CT Number)
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Syncytial Virus; Human Metapneumovirus
Keywords: mRNA-1345; mRNA-1365; RSV vaccine; hMPV vaccine; RSV/hMPV vaccine
MeSH Terms: interventions — mRNA-1345 respiratory syncytial virus vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Parts A and B are blinded, and Part C is open-label.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Part A: mRNA-1345, Dose 1 (Age Group: 8 to <24 months) (Experimental): Participants will receive mRNA-1345 vaccine by intramuscular (IM) injection on Days 1, 57 and 113.
  Interventions: Biological: mRNA-1345
- Part A: mRNA-1365, Dose 1 (Age Group: 8 to <24 months) (Experimental): Participants will receive mRNA-1365 vaccine by IM injection on Days 1, 57 and 113.
  Interventions: Biological: mRNA-1365
- Part A: Placebo (Age Group: 8 to <24 months) (Placebo Comparator): Participants will receive mRNA-1345/ mRNA-1365 vaccine matching placebo by IM injection on Days 1, 57 and 113. In countries where applicable, participants may receive Nimenrix instead of placebo on Day 113.
  Interventions: Biological: Placebo; Drug: Nimenrix
- Part B: mRNA-1345, Dose 2 (Age Group: 5 to <8 months) (Experimental): Participants will receive mRNA-1345 by IM injection on Days 1, 57 and 113.
  Interventions: Biological: mRNA-1345
- Part B: mRNA-1365, Dose 2 (Age Group: 5 to <8 months) (Experimental): Participants will receive mRNA-1365 by IM injection on Days 1, 57 and 113.
  Interventions: Biological: mRNA-1365
- Part B: mRNA-1345 Dose 1 (Age Group: 5 to <8 months) (Experimental): Participants will receive mRNA-1345 by IM injection on Days 1, 57 and 113.
  Interventions: Biological: mRNA-1345
- Part B: mRNA-1365 Dose 1 (Age Group: 5 to <8 months) (Experimental): Participants will receive mRNA-1365 by IM injection on Days 1, 57 and 113.
  Interventions: Biological: mRNA-1365
- Part B: Placebo (Age Group: 5 to <8 months) (Placebo Comparator): Participants will receive mRNA-1345/ mRNA-1365 vaccine matching placebo by IM injection on Days 1, 57 and 113. In countries where applicable, participants may receive Nimenrix instead of placebo on Day 113.
  Interventions: Biological: Placebo; Drug: Nimenrix
- Part C: mRNA-1345 Dose 1 (Age Group 8 to <12 months exposed to nirsevimab) (Experimental): Participants who have been previously exposed to nirsevimab will receive mRNA 1345 by IM on Days 1, 57, and 113.
  Interventions: Biological: mRNA-1345
- Part C: mRNA-1345 Dose 1 (Age Group 8 to <12 months not exposed to nirsevimab) (Experimental): Participants who have not been previously exposed to nirsevimab will receive mRNA 1345 by IM on Days 1, 57, and 113.
  Interventions: Biological: mRNA-1345

INTERVENTIONS:
Biological: mRNA-1345 — Sterile liquid for injection
  Arms: Part A: mRNA-1345, Dose 1 (Age Group: 8 to <24 months); Part B: mRNA-1345 Dose 1 (Age Group: 5 to <8 months); Part B: mRNA-1345, Dose 2 (Age Group: 5 to <8 months); Part C: mRNA-1345 Dose 1 (Age Group 8 to <12 months exposed to nirsevimab); Part C: mRNA-1345 Dose 1 (Age Group 8 to <12 months not exposed to nirsevimab)
Biological: mRNA-1365 — Sterile liquid for injection
  Arms: Part A: mRNA-1365, Dose 1 (Age Group: 8 to <24 months); Part B: mRNA-1365 Dose 1 (Age Group: 5 to <8 months); Part B: mRNA-1365, Dose 2 (Age Group: 5 to <8 months)
Biological: Placebo — 0.9% sodium chloride (normal saline) solution for injection
  Arms: Part A: Placebo (Age Group: 8 to <24 months); Part B: Placebo (Age Group: 5 to <8 months)
Drug: Nimenrix — Solution for injection
  Arms: Part A: Placebo (Age Group: 8 to <24 months); Part B: Placebo (Age Group: 5 to <8 months)

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of mRNA-1365, an mRNA vaccine targeting respiratory syncytial virus (RSV) and human metapneumovirus (hMPV) and mRNA-1345, an mRNA vaccine targeting RSV, in participants aged 5 months to <24 months.

ELIGIBILITY:
Inclusion Criteria:

* The participant is 8 months to <24 months (Part A), 5 months to <8 months (Part B), or 8 months to <12 months (Part C) of age at the time of randomization (Day 1/Baseline visit), who is in good general health, in the opinion of the Investigator, based on review of medical history and screening physical examination.
* In the Investigator's opinion, the parent(s)/ legally authorized representative (LAR)(s) understand and are willing and physically able to comply with protocol-mandated follow up, including all procedures, and provide written informed consent.
* The participant is growing normally for age in the opinion of the site clinician in the months prior to enrollment.
* The participant was born at full-term (≥37 weeks gestation) with a minimum birth weight of 2.5 kilograms (kg).
* For Part C Cohort 7: participant must have received nirsevimab ≥6 months prior to Day 1 Visit.
* For Part C Cohort 8: participant was eligible at any time since birth, according to national guidelines, to receive nirsevimab prior to Day 1 Visit but did not do so.

Exclusion Criteria:

* Has a known history of symptomatic RSV (Part A: within 3 months; Part B and Part C: since birth) or hMPV infection (Part A: within 3 months; Part B: since birth) prior to administration of the first dose of investigational product (IP) or has a known close contact with anyone with laboratory-confirmed RSV (Parts A, B, and C) or hMPV infection (Parts A or B) within 14 days prior to administration of the first dose of IP.
* Is acutely ill or febrile 24 hours prior to or at the screening visit. Fever is defined as a body temperature ≥38.0°Celsius/≥100.4°Fahrenheit. Participants who meet this criterion may have visits rescheduled within the relevant study visit windows.
* Has previously been administered an investigational or approved vaccine for prevention of RSV (Parts A, B, and C) or hMPV (Parts A and B) infection or if the participant's mother received an investigational or approved vaccine for the prevention of RSV (Parts A, B, and C) or hMPV (Parts A and B) infection during pregnancy.
* Has received investigational or approved agents for prophylaxis against RSV or hMPV (for example, monoclonal antibodies) or is intending to receive these during the course of the study. For Part C (Cohort 7 only), use of nirsevimab ≥6 months before Day 1 Visit is allowed.
* Has a known hypersensitivity to a component of the vaccine or its excipients. Hypersensitivity includes, but is not limited to, anaphylaxis or immediate allergic reaction of any severity to a previous dose of an mRNA vaccine or any of its components (including polyethylene glycol or immediate allergic reaction of any severity to polysorbate).
* Has a medical condition that, according to the Investigator's judgment, may pose additional risk as a result of participation, interfere with safety assessments, or interfere with interpretation of results.

Note: Other protocol-defined inclusion/exclusion criteria apply.

Ages: 5 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 186 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local and Systemic Adverse Reactions (ARs) | Up to Day 120 (7 days after each injection)
Number of Participants with Unsolicited Adverse Events (AEs) | Up to Day 141 (28 days after each injection)
Number of Participants with Medically-Attended Adverse Events (MAAEs) | Day 1 through Day 730
Number of Participants with Adverse Event of Special Interests (AESIs), Serious Adverse Events (SAEs) and Adverse Events Leading to Discontinuation | Day 1 through Day 730

SECONDARY OUTCOMES:
Number of Participants with Respiratory Tract Illness (RTI), Lower Respiratory Tract Illness (LRTI), Severe LRTI, Very Severe LRTI, and Hospitalizations Associated with RSV or hMPV | Day 1 through Day 730
Parts A and B: Geometric Mean Titer (GMT) of Serum RSV and hMPV Neutralizing Antibodies | Baseline up to Month 12
Part C: GMT of Serum RSV Neutralizing Antibodies | Baseline up to Month 12
Parts A and B: Geometric Mean Concentration (GMC) of Serum RSV F- and hMPV F-Binding Antibodies | Baseline up to Month 12
Part C: GMC of Serum RSV F-Binding Antibodies | Baseline up to Month 12
Geometric Mean Fold-Rise (GMFR) Postbaseline/baseline Neutralizing Antibody Titers | Baseline up to Month 12
Number of Participants with Vaccine-specific T-cell Responses Measured by Flow Cytometry | Baseline up to month 12

CONTACTS AND LOCATIONS:
Locations (49):
- United States (29):
  - Matrix Clinical Research, Los Angeles, California
  - Los Angeles Children's Hospital, Los Angeles, California
  - Velocity Clinical Research, Denver, Englewood, Colorado
  - Meridian Clinical Research, Washington D.C., District of Columbia
  - University Of Florida Health Science Center, Jacksonville, Florida
  - Accel Research Sites - Nona Pediatric Center, Orlando, Florida
  - Clinical Research Prime, Idaho Falls, Idaho
  - MedPharmics - Platinum - PPDS, Lafayette, Louisiana
  - Umass Memorial Medical Center, Worcester, Massachusetts
  - UMASS Chan Medical School, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Great Lakes Research Institute, Southfield, Michigan
  - Pediatric Specialty Care Discovery Clinic, Minneapolis, Minnesota
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Meridian Clinical Research, Hastings, Nebraska
  - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Senders Pediatrics, South Euclid, Ohio
  - Velocity Clinical Research - Providence, Providence, Rhode Island
  - Palmetto Pediatrics, PA, North Charleston, South Carolina
  - Vanderbilt Vaccine Research Program, Nashville, Tennessee
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Mercury Clinical Research, Inc., Houston, Texas
  - CyFair, Houston, Texas
  - Pediatric Associates, Houston, Texas
  - Village Pediatrics, Plano, Texas
  - Mercury Clinical Research, Inc., Richmond, Texas
  - Pediatric Center, Richmond, Texas
  - North Houston Internal Medicine & Pediatric Clinic, Tomball, Texas
  - Childrens Hospital Regional Medical Center, Seattle, Washington
- Telethon Kids Institute, Nedlands, Western Australia, Australia
- Canada (4):
  - BC Children's Hospital - Vaccine Evaluation Centre - Neonatology, Vancouver, British Columbia
  - Dalhousie University IWK Health Centre, Halifax, Nova Scotia
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - Universite de Montreal - Centre Hospitalier Universitaire (CHU) Sainte-Justine, Montreal, Quebec
- Panama (4):
  - CEVAXIN David, David, Chiriquí Province
  - CEVAXIN Chorrera, La Chorrera, Panamá Oeste Province
  - CEVAXIN Avenida Mexico, Panama City
  - CEVAXIN 24 de Diciembre, Panama City
- South Africa (5):
  - Shandukani Research CRS, Hillbrow, Gauteng
  - Wits Health Consortium, Johannesburg, Gauteng
  - Setshaba Research centre, Soshanguve, Gauteng
  - Family Centre for Research with Ubuntu (FAMCRU)- Tygerberg, Cape Town, Western Cape
  - Practice Dr Jan Vermeulen, Cape Town, Western Cape
- United Kingdom (6):
  - Alder Hey NHS Foundation Trust - Pharmacy Clinical Trials, Liverpool
  - St George's Hospital, London
  - Imperial College London and Imperial College Healthcare NHS, London
  - Norfolk and Norwich University Hospitals, Norwich
  - John Radcliffe Hospital, Oxford
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Amodio D, Angelidou A, Cotugno N, Sherman AC, Levy O, Palma P; IPVC 2023 Speakers' group. Biomarkers of vaccine safety and efficacy in vulnerable populations: Lessons from the fourth international precision vaccines conference. Vaccine. 2025 Jan 1;43(Pt 2):126477. doi: 10.1016/j.vaccine.2024.126477. Epub 2024 Nov 28. PMID 39608233